CLINICAL TRIAL: NCT01603290
Title: Change of Fatigue and Physical Fitness and Their Related Factors in Hospitalized Hematology Patients
Brief Title: Change of Fatigue and Physical Fitness in Hospitalized Hematology Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Institutional Review Board, National Taiwan University Hospital
Other Study IDs: 201111066RIC
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Acute Leukemia
Keywords: Acute leukemia,; Chemotherapy,; Cancer-Related Fatigue,; Physical Fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hospitalized Leukemia Patients: leukemia patients with chemotherapy during hospitalization

SUMMARY:
The purposes of this study are to (1) explore the severity of symptom of leukemia patients experienced before and after chemotherapy in hospital, (2) investigate the trajectories of the fatigue and physical fitness, and their related factors, and (3) the correlation between fatigue and physical fitness

DETAILED DESCRIPTION:
Cancer-Related Fatigue (CRF) is one of the common distressed symptoms that leukemia patients experienced during the period of chemotherapy. Exercise is the most effective non-pharmacologic treatment but inpatients refuse to do exercise in clinical settings in Taiwan. Decreased physical activity may increase the intensity of fatigue and degenerate the physical fitness; however, there is no study to explore the trajectories of fatigue and physical fitness for leukemia patient during hospitalization. Therefore, the purposes of this study are to (1) explore the severity of symptom of leukemia patients experienced before and after chemotherapy in hospital, (2) investigate the trajectories of the fatigue and physical fitness, and their related factors, and (3) the correlation between fatigue and physical fitness. A longitudinal designed study will be conducted to recruit the leukemia patients in a medical center in Taipei. Eligible patients are those will be going to receive chemotherapy and in hospital at least one week. Time periods for data collection will be in the first 48 hours after hospitalization (T0) and the 48 hours before the patient discharged (T1). A set of structured questionnaire will be used to collected data including the Background information form, the Fatigue Symptom Inventory, the Cancer Fatigue Scale, the Symptom Severity Scale, and the Hospital Anxiety and Depression Scale. Patients will be received physical fitness test including the 6-Minute Walking Test, grip strength, and 30-second chair stand test. The descriptive statistics will be used to analyze the severity of symptom distress, fatigue, and the change of physical fitness, and the inferential statistics was used to analyze the correlation of the symptom, fatigue, and physical fitness. Besides, generalized estimating equations (GEE) will be used to analysis the average of population change of fatigue and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Acute leukemia patients with first complete remission status
* Aged above 20
* Be going to receive chemotherapy and in hospital at least one week.
* Those Who willing to participate in the research

Exclusion Criteria:

* Physician consider the patient was not suitable
* Patients' limbs can not move
* Patients' conscious was unclear during hospitalization
* Patient with pain of joint and can't do 30-second chair stand test and 6-Minute Walking Test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute leukemia inpatients
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan